CLINICAL TRIAL: NCT05898230
Title: Retrospective Clinical Data Collection on Carbomedics OptiForm Mitral Heart Valve
Status: Recruiting | Type: Observational
Sponsor: Corcym S.r.l (Industry)
Responsible Party: Sponsor
Other Study IDs: CCH802
Record Dates: First submitted 2023-06-01; First posted 2023-06-12 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Mitral Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subjects who have been implanted with the Carbomedics OptiForm Mitral Heart Valve: Mitral Valve Replacement with Carbomedics OptiForm Mitral Heart Valve
  Interventions: Device: Mitral Valve Replacement

INTERVENTIONS:
Device: Mitral Valve Replacement — Mitral Valve Replacement with Carbomedics OptiForm Mitral Heart Valve

SUMMARY:
The objective of this study is to evaluate the medium- to long-term safety of the Carbomedics OptiForm Mitral Heart Valve after the implantation for mitral valve disease in the Chinese population.

The study is designed as a post-market, retrospective, single arm and multicentric data collection

DETAILED DESCRIPTION:
This study is conducted to evaluate the medium and long-term safety of the Carbomedics OptiForm Mitral Heart Valve after the implantation for mitral valve disease. The data will be used for regulatory purposes, to support the re-certification of the valve in the Chinese market.

Valve-related SAEs such as prosthetic valve dysfunction, death, valve-related bleeding events, valve thrombosis and thromboembolic events, endocarditis and reintervention will be studied to describe the safety profile of the valve. Data of approximately 400 subjects will be collected in two clinical sites in China.

ELIGIBILITY:
Inclusion Criteria:

* Subject who has been treated with the Carbomedics OptiForm Mitral Heart Valve.
* Subject (or representative or family member) who can understand the objective of the study and is willing to provide verbal informed consent and the available medical information.

Exclusion Criteria:

* Subject (or legal representative or family member) who do not provide their verbal consent to the data collection, or who are unable to provide follow-up information

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who have been implanted with the Carbomedics OptiForm Mitral Heart Valve
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Prosthetic Valve Dysfunction | up to 7-8 year
  The number and percentage of subjects with Prosthetic valve Dysfuntion
Mortality | up to 7-8 year
  The number and percentage of subjects died
Valve-related bleeding | up to 7-8 year
  The number and percentage of subjects with Valve-related bleeding
Valve thrombosis | up to 7-8 year
  The number and percentage of subjects with Valve Thrombosis
Thromboembolism | up to 7-8 year
  The number and percentage of subjects with Thromboembolic events
Endocarditis | up to 7-8 year
  The number and percentage of subjects with Endocarditis
Valve-Related Reintervention | up to 7-8 year
  The number and percentage of subjects underwent Valve-related reintervention

CONTACTS AND LOCATIONS:
Overall Officials: Sara Gaggianesi, Study Director — Corcym S.r.l
Locations (2):
- China (2):
  - The second Xiangya Hospital of Central South University, Changsha
  - West China hospital of Sichuan University, Chendu